CLINICAL TRIAL: NCT01126645
Title: Evaluation of Sorafenib in Combination With Local Micro-therapy Guided by Gd-EOB-DTPA Enhanced MRI in Patients With Inoperable Hepatocellular Carcinoma
Brief Title: Sorafenib and Micro-therapy Guided by Primovist Enhanced MRI in Patients With Inoperable Liver Cancer
Acronym: SORAMIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: Bayer (Industry); Sirtex Medical (Industry)
Responsible Party: Principal Investigator, Jens Ricke, Prof. Dr. Jens Ricke, University Hospital Munich, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT No. 2009-012576-27
Record Dates: First submitted 2010-05-17; First posted 2010-05-20 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Sirtuins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- local ablation group (Other): Local ablation group: Potentially curative treatment of early HCC includes surgical resection and local ablation (RFA, PEI, BT). Recurrence rates after such approaches are reported to amount to 50% at 3 years and 70% at 5 years. Tumor recurrence may be either due to de novo development of new primary tumors or due to intrahepatic (unrecognized) metastases. Prevention of recurrence after local ablation is an important strategy to improve overall survival. So far, adjuvant chemoembolization and chemotherapy have not proven to be effective in preventing recurrences. There is, however, a strong rationale to assume that sorafenib will be of value in the adjuvant treatment of HCC as sorafenib has a dual mechanism of action (inhibition of tumor proliferation and antiangiogenesis) and has proven efficacy in HCC.
  Interventions: Procedure: RFA
- palliative treatment group (Active Comparator): Radioembolization has been reported to be effective in patients with unresectable HCC with preserved liver function from a number of trials. Successful downstaging of disease rendering patients eligible for potentially curative therapies, and even histologically confirmed complete responses of unresectable HCC, have repeatedly been reported providing the rationale to evaluate SIRT+sorafenib in comparison to sorafenib alone.
  The impact of cirrhosis as a concomitant disease in most patients with HCC is that it limits the ability of many patients to tolerate chemotherapy and is an independent cause of death in HCC patients. Thus, the historical difficulty in demonstrating an effect of therapy on survival in patients with advanced-stage, unresectable HCC (the majority). A new therapy that is effective in controlling hepatic disease, is less toxic than traditional chemotherapy, and improves the quality of life for patients in the advanced stages of HCC could represent an alternative.
  Interventions: Procedure: Radioembolization (SIRT)

INTERVENTIONS:
Procedure: RFA — A max.of 2 percutaneous RFA sessions is permitted per patient with a max.of 2 liver lesions treated in each RFA session. Randomization to sorafenib or placebo is performed after completion of RFA. Percutaneous RFA is to be performed according to the manufacturer's instructions and following as far as possible routine procedures of the participating hospital. Typically, RFA will be performed under conscious sedation, general anesthesia is permitted. After local anesthesia of the site of puncture, the applicator is positioned in the center of the lesion using ultrasound-, CT- or MR-guidance. The success of ablation is to be controlled directly after RFA using ultrasound, contrast-enhanced CT, or MR imaging. If for any reason RFA is deemed incomplete within the immediate follow-up (up to 2 weeks after the initial ablation), RFA is to be repeated once (in this case, the total (max.) number of RFA sessions will be three).
  The study procedure guide will contain further instructions for RFA.
  Other Names: Sorafenib (Nexavar 200 mg film-coated tablets),marketing authorization no.:EU/1/06/342/001
  Arms: local ablation group
Procedure: Radioembolization (SIRT) — One SIRT prescription consists of the pre-treatment assessment followed by one or 2 treatment sessions The aim of pre-treatment assessment is to ensure delivery of the microspheres to the target. Evaluation includes a determination of the arterial location and any consequent necessity for coil-embolization of the gastroduodenal artery, right gastric artery and any other accessory arteries to prevent inadvertent administration of microspheres into the gastrointestinal tract or pancreas. In addition, parasitic extrahepatic supply should be coil-embolized.
  Patients in whom the shunt fraction indicates potential exposure to the lung to an absorbed radiation dose of more than 30 Gy should be excluded from treatment with SIR-Spheres. Patients who are randomized to receive SIRT but who are not regarded as eligible for SIRT after the pre-treatment assessment will be switched to the sorafenib only group within the palliative treatment arm.
  Other Names: SIR Spheres Microspheres; Sorafenib (Nexavar)
  Arms: palliative treatment group

SUMMARY:
The purpose of this study is to evaluate Sorafenib and local microtherapy guided by Primovist enhanced MRI in patients with inoperable liver cancer (HCC).

Methodology:

Patients with a diagnosis of hepatocellular carcinoma will receive either:

* local ablation therapy of liver lesions by radiofrequency ablation followed by sorafenib or placebo (local ablation group), or
* radioembolization (SIRT) + sorafenib or sorafenib alone (palliative treatment group).

In each study group, patients will be randomized to one of the two treatment arms following a pre-defined randomization plan. Randomization will be on a 1:1 basis in the local ablation group and on the basis of 10 (sorafenib only) : 11 (SIRT + sorafenib) in the palliative treatment group.

Patients in the local ablation group will be followed at 2 months intervals for recurrence and overall survival, patients in the palliative treatment group will be followed for overall survival. Follow-up in each study group will end 24 months after inclusion of the last patient into the respective study group.

The assignment of patients to the local ablation or palliative study group will be based on the ablative potential of RFA (local ablation if ≤4 tumors, each ≤5 cm in size). Diagnostic imaging will be used to guide this decision. The assignment to the local ablation or the palliative treatment group will be made by the local investigator.

As a sub-study, all patients will undergo Primovist®-enhanced MRI in addition to contrast-enhanced CT before assignment to one treatment group. The goal of the sub-study is to assess the value of Primovist®-enhanced MRI to correctly stratify patients for a local ablation or palliative treatment strategy. Primovist®-enhanced MRI will be compared with contrast-enhanced multislice CT using a truth panel assessment as the standard of reference. In addition, Primovist-enhanced MRI and contrast-enhanced CT will be obtained during follow-up of patients in the local ablation group to assess its potential for detection of recurrence.

ELIGIBILITY:
Inclusion Criteria

1. Age: 18-85 years
2. Diagnosis of hepatocellular carcinoma
3. If primary diagnosis of HCC: diagnosis based on the following criteria:

   1. cyto-histological criteria, OR
   2. radiological criteria: Focal lesion >1 cm with arterial hypervascularization in 2 coincident imaging techniques (CT, MRI, or US), OR
   3. combined criteria: one imaging technique showing a focal lesion 1-2 cm with arterial hypervascularization AND AFP levels >400 ng/mL, OR
   4. combined criteria: one imaging technique showing a focal lesion >2 cm with arterial hypervascularization AND AFP levels >200 ng/mL
4. If extrahepatic metastases: liver-dominant disease
5. Stage BCLC A, B, or C
6. Child-Pugh A, Child-Pugh B up to 7 points (in patients receiving anticoagulant therapy: Child-Pugh score up to 5 points; INR category not regarded for calculation of the Child-Pugh score)
7. Willing to comply with all study procedures
8. Has voluntarily given written informed consent

Exclusion Criteria

1. If female, pregnant or breast feeding (females of child-bearing potential must use adequate contraception and must have a negative pregnancy test performed within 7 days prior to inclusion into this study)
2. If male, not using adequate birth control measures
3. One or more of the following:

   * Hemoglobin <10g/dL,
   * WBC <2,500 cells/mm3,
   * ANC <1,500 cells/mm3,
   * platelets <50,000/mm3,
   * ECOG performance status >2
4. Life expectancy <16 weeks or medically unstable
5. Extrahepatic metastases (except metastases to bone, lymph nodes, and adrenal glands which do not constitute an exclusion criterion), but, see Additional Criteria for the Local Ablation Group, below (Section 4.2 of the study protocol)
6. Patients with known GFR <30 mL/min/1.73m2
7. PT-INR/PTT >1.5 times the upper limit of normal (patients on anticoagulation therapy will be allowed to participate provided that no prior evidence exists of an underlying abnormality in anticoagulation)
8. Uncontrolled infections at the time of microtherapy
9. Child-Pugh score >7 points; in patients receiving anticoagulant therapy: Child-Pugh score >5 points (INR category not regarded for calculation of the Child-Pugh score)
10. Uncontrolled ascites
11. Tumor load of the whole liver >70%
12. Contraindications for study medications according to product labeling or procedures (sorafenib, Primovist®, x-ray contrast agents, SIR-Spheres®, RFA, MWA, MRI, CT) incl. any contraindication to the transarterial interventional procedure (e.g., allergy against x-ray contrast agents, uncontrolled hyperthyroidism)
13. Prior resection of the papilla of Vater (e.g., Whipple procedure) or bile duct stent across the papilla
14. Significant cardiovascular disease; e.g., myocardial infarction within 6 months of inclusion, chronic heart failure (New York Heart Association class III or IV), unstable coronary artery disease
15. Uncontrolled hypertension
16. Thrombotic or embolic events including transient ischemic attacks within the past 6 months (tumor-related portal vein thrombosis allowed in the palliative part of the trial).
17. History of GI bleeding within 30 days before inclusion into this study
18. History of esophageal varices bleeding which has not been controlled by effective therapy and/or therapy to prevent bleeding recurrence
19. Previous malignancy other than carcinoma in situ of the skin or the cervix uteri within 5 years prior to inclusion
20. History of organ transplant (including prior liver transplantation)
21. HIV, congenital immune defect, any immunosuppressive therapy for autoimmune disease (rheumatoid arthritis) or inflammatory bowel disease
22. Mental conditions rendering the subject incapable to understand the nature, scope, and consequences of the trial
23. Close affiliation with the investigational site; e.g. first-degree relative of the investigator
24. Participating in another therapeutic clinical trial or has completed study participation in another therapeutic clinical trial within 30 days of enrolment into this trial
25. Having been previously enrolled in this clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
time to recurrence | 13-18 months (average time to recurrence)
  In patients in whom local ablation therapy is appropriate, to determine if the sorafenib in combination with radiofrequency ablation (RFA) prolongs the time-to-recurrence (TTR) in comparison with RFA + placebo.
overall survival | 10-15 months (average survival)
  In patients in whom RFA is NOT appropriate (palliative treatment group), to determine if the combination of yttrium-90 microspheres (SIRT) + sorafenib improves the overall survival (OS) in comparison to sorafenib alone.
  Interim analysis will be conducted after 60 and 180 deaths and a final analysis after 240 deaths.
Primovist®-enhanced MRI is non-inferior or superior compared with contrast-enhanced multislice CT | 3 years
  To confirm in a 2-step procedure that Primovist®-enhanced MRI is non-inferior (first step) or superior (second step) compared with contrast-enhanced multislice CT for assignment of patients to a palliative vs. local ablation treatment strategy.
  The overall study is successful, if the primary objectives 1 OR 2 are met, AND Primovist-enhanced MRI is at least non-inferior to contrast-enhanced CT for treatment stratification.

SECONDARY OUTCOMES:
quality of life | 3 years
  assess health-related quality of life via ECOG questionnaire
safety of RFA | 3 years
  To assess the safety of the combination of RFA + sorafenib in comparison to RFA + placebo
safety of SIR Spheres | 3 years
  To assess the safety of the combination of SIR-Spheres therapy and sorafenib in comparison to sorafenib alone.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ricke, Prof. Dr., Study Director — University Hospital Munich; Peter Malfertheiner, Prof. Dr., Study Director — University of Magdeburg
Locations (1):
- University of Magdeburg, Magdeburg, Germany

REFERENCES:
- [Derived] Seidensticker M, Ocal O, Schutte K, Malfertheiner P, Berg T, Loewe C, Klumpen HJ, van Delden O, Umutlu MR, Ben Khaled N, de Toni EN, Seidensticker R, Aghdassi A, Tran A, Bronowicki JP, Peynircioglu B, Sangro B, Pech M, Ricke J. Impact of adjuvant sorafenib treatment after local ablation for HCC in the phase II SORAMIC trial. JHEP Rep. 2023 Feb 15;5(5):100699. doi: 10.1016/j.jhepr.2023.100699. eCollection 2023 May. PMID 36968218
- [Derived] Ricke J, Schinner R, Seidensticker M, Gasbarrini A, van Delden OM, Amthauer H, Peynircioglu B, Bargellini I, Iezzi R, De Toni EN, Malfertheiner P, Pech M, Sangro B. Liver function after combined selective internal radiation therapy or sorafenib monotherapy in advanced hepatocellular carcinoma. J Hepatol. 2021 Dec;75(6):1387-1396. doi: 10.1016/j.jhep.2021.07.037. Epub 2021 Aug 27. PMID 34454995
- See also: web page of SORAMIC clinical trial — http://www.soramic.com